CLINICAL TRIAL: NCT00810472
Title: Clinical Trial to Investigate Superiority of HLA Matching in Comparison to Random Graft Assignment With Respect to the Endpoint 'Time to First Endothelial Graft Rejection' in Penetrating Keratoplasty.
Brief Title: Functional Antigen Matching in Corneal Transplantation
Acronym: FANCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Daniel Böhringer, Apl.Prof.Dr.med., University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FR-2008-FANCY
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Corneal Diseases
Keywords: Penetrating keratoplasty; HLA matching; Corneal diseases that require penetrating keratoplasty
MeSH Terms: conditions — Corneal Diseases | interventions — Keratoplasty, Penetrating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HLA Matching (Experimental): HLA matching is exerted by selecting the donor with least-most additional HLA alleles. We will predict the waiting time for such a donor in order to assess eligibility for the trial [8]. In addition, we will dynamically adopt the degree of matching that is aimed at depending on the predicted time interval and actual waiting time: the first donors not exerting more than 7 mismatches at the triplet-amino-acid-residue-level (HLAMatchmaker method [6]) is accepted if the patient is waiting less than half of his predicted waiting time. The next available donor exerting a 2/6 match (or better) is assigned thereafter. The next graft will be assigned, regardless of HLA matching after 6 months.
  Interventions: Other: HLA Matching; Procedure: Penetrating keratoplasty
- Random graft assignment (Placebo Comparator)
  Interventions: Procedure: Penetrating keratoplasty

INTERVENTIONS:
Other: HLA Matching — HLA matching is exerted by selecting the donor with least-most additional HLA alleles. We will predict the waiting time for such a donor in order to assess eligibility for the trial [8]. In addition, we will dynamically adopt the degree of matching that is aimed at depending on the predicted time interval and actual waiting time: the first donors not exerting more than 7 mismatches at the triplet-amino-acid-residue-level (HLAMatchmaker method [6]) is accepted if the patient is waiting less than half of his predicted waiting time. The next available donor exerting a 2/6 match (or better) is assigned thereafter. The next graft will be assigned, regardless of HLA matching after 6 months.
  Arms: HLA Matching
Procedure: Penetrating keratoplasty — Corneal transplantation.

SUMMARY:
Penetrating keratoplasty is one of the most commonly performed transplantation surgeries. Graft rejection is a major complication. HLA compatibility has already been demonstrated an effective prophylaxis in several retrospective investigations. The purpose of the investigators randomized clinical trial is to demonstrate superiority of HLA matching in comparison to random graft assignment with respect to the endpoint 'time to first endothelial graft rejection' in penetrating keratoplasty. The investigators will perform DNA-based allele resolution typing.

ELIGIBILITY:
Inclusion Criteria:

* Predicted waiting time for a 4/6 match lower than 6 months.

Exclusion Criteria:

* Minority
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2009-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time to first endothelial graft rejection. | Mostly within the first six months.

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Bohringer D, Spierings E, Enczmann J, Bohringer S, Sundmacher R, Goulmy E, Reinhard T. Matching of the minor histocompatibility antigen HLA-A1/H-Y may improve prognosis in corneal transplantation. Transplantation. 2006 Oct 27;82(8):1037-41. doi: 10.1097/01.tp.0000235908.54766.44. PMID 17060851
- [Background] Reinhard T, Spelsberg H, Henke L, Kontopoulos T, Enczmann J, Wernet P, Berschick P, Sundmacher R, Bohringer D. Long-term results of allogeneic penetrating limbo-keratoplasty in total limbal stem cell deficiency. Ophthalmology. 2004 Apr;111(4):775-82. doi: 10.1016/j.ophtha.2003.07.013. PMID 15051212
- [Background] Reinhard T, Bohringer D, Enczmann J, Kogler G, Mayweg S, Wernet P, Sundmacher R. Improvement of graft prognosis in penetrating normal-risk keratoplasty by HLA class I and II matching. Eye (Lond). 2004 Mar;18(3):269-77. doi: 10.1038/sj.eye.6700636. PMID 15004576
- [Background] Bohringer D, Reinhard T, Duquesnoy RJ, Bohringer S, Enczmann J, Lange P, Claas F, Sundmacher R. Beneficial effect of matching at the HLA-A and -B amino-acid triplet level on rejection-free clear graft survival in penetrating keratoplasty. Transplantation. 2004 Feb 15;77(3):417-21. doi: 10.1097/01.TP.0000110415.10401.94. PMID 14966417
- [Background] Reinhard T, Bohringer D, Enczmann J, Kogler G, Wernet P, Bohringer S, Sundmacher R. HLA class I/II matching and chronic endothelial cell loss in penetrating normal risk keratoplasty. Acta Ophthalmol Scand. 2004 Feb;82(1):13-8. doi: 10.1046/j.1600-0420.2003.00188.x. PMID 14738484
- [Background] Bohringer D, Reinhard T, Enczmann J, Godehard E, Sundmacher R. Individual analysis of expected time on the waiting list for HLA-matched corneal grafts. Dev Ophthalmol. 2003;36:50-5. doi: 10.1159/000067648. PMID 12494680
- [Derived] Bohringer D, Grotejohann B, Ihorst G, Reinshagen H, Spierings E, Reinhard T. Rejection Prophylaxis in Corneal Transplant. Dtsch Arztebl Int. 2018 Apr 13;115(15):259-265. doi: 10.3238/arztebl.2018.0259. PMID 29735006
- [Derived] Bohringer D, Ihorst G, Grotejohann B, Maurer J, Spierings E, Reinhard T; FANCY study group. Functional antigen matching in corneal transplantation: matching for the HLA-A, -B and -DRB1 antigens (FANCY) - study protocol. BMC Ophthalmol. 2014 Dec 13;14:156. doi: 10.1186/1471-2415-14-156. PMID 25496165